CLINICAL TRIAL: NCT02582892
Title: Systemic Vitamin D Supplementation in Menopausal Women With Dental Implants
Brief Title: Systemic Vitamin D Supplementation in Dental Implants Patients
Acronym: VitaminD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Potiguar (Other)
Responsible Party: Principal Investigator, MARCO BOTELHO, Program Director of Graduate Biotechnology, University Potiguar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVIDENCE x UNP VITAMIN D
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vit D (Other): Vit D 20 mg/day
  Interventions: Drug: Vit D

INTERVENTIONS:
Drug: Vit D — 20 mg/day
  Other Names: Vitamin D

SUMMARY:
Vitamin D plays an essential role in calcium homeostasis and is critical for bone formation and remodeling.

DETAILED DESCRIPTION:
Evidence has demonstrated that vitamin D deficiency plays an important role in dental implants outcomes.

Low serum levels of Vitamin D is considered as a risk factor, not only for low mineral bone density but also in other metabolic pathways such as those involved in immune response and chronic inflammatory diseases.

There are few studies demonstrating the role that vitamin D deficiency in the etiopathogenesis of oral diseases and the consequences in Dental Implants.

Dentists have not yet well understood the importance of a good bone metabolism response for a successful bone regeneration and osseointegration of implants.

An insufficient bone response can not guarantee the necessary stability of the implants placed in it, has been one of the biggest problems of implantology.

Thus, the aim of this study is to evaluate the efficacy of Systemic vitamin D supplementation in menopausal women cadidates for dental implants.

ELIGIBILITY:
Inclusion Criteria:

- Menopause patients

Exclusion Criteria:

* patients with a past history of neurological disorder;
* who had received pharmacotherapy for depression within 8 weeks of screening;
* who were taking medication known to interfere with Vit D;
* who had recent psychiatricor systemic illness;
* uncontrolled hypertension (blood pressure > 160/95mmHg);
* unstable cardiovascular disease;
* User of psychoactive medications;
* alcohol excess consumption abuse.

Ages: 3 Months to 5 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
25 OH Serum levels | 2 years
  VIT D Serum levels

SECONDARY OUTCOMES:
Osteoporosis condition | 2 years
  Densitometry in patients femur bones

CONTACTS AND LOCATIONS:
Overall Officials: Gugliemo G Campus, PhD, Study Chair — Università degli Studi di Sassari
Locations (3):
- Brazil (3):
  - Gynelogical Center, Fortaleza, Ceará
  - University Potiguar, Natal, Rio Grande do Norte
  - Marco Botelho, São Paulo, São Paulo

REFERENCES:
- [Result] Botelho MA, Queiroz DB, Barros G, Guerreiro S, Fechine P, Umbelino S, Lyra A, Borges B, Freitas A, Queiroz DC, Ruela R, Almeida JG, Quintans L Jr. Nanostructured transdermal hormone replacement therapy for relieving menopausal symptoms: a confocal Raman spectroscopy study. Clinics (Sao Paulo). 2014 Feb;69(2):75-82. doi: 10.6061/clinics/2014(02)01. PMID 24519196
- [Result] Botelho MA, Martins JG, Ruela RS, Queiroz DB, Ruela WS. Nanotechnology in ligature-induced periodontitis: protective effect of a doxycycline gel with nanoparticules. J Appl Oral Sci. 2010 Jul-Aug;18(4):335-42. doi: 10.1590/s1678-77572010000400003. PMID 20835566